CLINICAL TRIAL: NCT00669435
Title: Ultrasonographic Modification of Liver Steatosis and Visceral Fat Induced by Treatment With Losartan and Simvastatin in Hypertensive Normocholesterolemic Obese Patients
Brief Title: Losartan and Simvastatin in Hypertensive Obeses With Liver Steatosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pavia (Other)
Responsible Party: Giuseppe Derosa/MD, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIPV003DIM2008
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: Essential hypertension; Liver steatosis
MeSH Terms: conditions — Hypertension; Essential Hypertension; Fatty Liver | interventions — Losartan; Simvastatin; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Amlodipine and Simvastatin
  Interventions: Drug: Amlodipine + Simvastatin
- 2 (Experimental): Losartan and Simvastatin
  Interventions: Drug: Losartan + Simvastatin

INTERVENTIONS:
Drug: Losartan + Simvastatin — tablets; 50, 100 mg; od; 12 months
  tablets; 20 mg; od; 6 months
  Arms: 2
Drug: Amlodipine + Simvastatin — tablets; 5, 10 mg; od; 12 months
  tablets; 20 mg; od; 6 months
  Arms: 1

SUMMARY:
Angiotensin II has been proposed as a lipid metabolism regulator. It is known that adipocytes secrete a variety of protein, such as TNFα, plasminogen activator inhibitor (PAI)-1, leptin, resistin and adiponectin; these proteins have a wide range of biological effects and are associated with insulin resistance. Adipocytes also produce angiotensinogen and angiotensin II and a local renin-angiotensin system (RAS) is present in adipose tissue. In overweight or obese hypertensive normocholesterolemic patients the treatment with AT1-receptor blocker (Losartan) may have a better effect on hepatic steatosis and visceral fat deposition than the antihypertensive treatment with calcium channel blocker (amlodipine). Simvastatin will be added to both groups. The aim of this study is to evaluate the effect of losartan and simvastatin on ultrasonographic qualitative and quantitative parameters in overweight or obese hypertensive normocholesterolemic patients with hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Gender: 50% Male and 50% female
* Age: 40-80 years
* Race: Caucasian
* Overweight or obese: respectively BMI25-30 kg/m2 or BMI > 30 kg m2
* Hypertensive: PA > 140/90 mmHg
* Normocholesterolemic (LDL< 160 mg/dl HDL > 35 mg/dl)
* Liver steatosis

Exclusion Criteria:

* other antihypertensive treatment after wash out period of 2 weeks
* abnormal heart rest function (EF < 55%).
* valvular heart disease
* congenital heart disease
* heart failure or prior myocardial infarction
* diabetes
* renal disease
* liver disease
* connective tissue disease
* pregnancy or lactation
* serious adverse experience
* sensitivity to the study drugs or its components
* contraindication from an approved label

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
All patients will undergo anthropometric evaluation and abdominal ultrasonography (performed by the same examiner); will be taken routine liver US and US measurement of visceral and subcutaneous fat. | Between 08.00 and 10.00 at baseline, and after 1, 6, and 12 months

SECONDARY OUTCOMES:
Determination of insulin sensitivity, leptin, adiponectin, TNFα, IL6, hsPCR | Between 08.00 and 10.00 at baseline, and after 1, 6, and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pavia, Pavia, Italy